CLINICAL TRIAL: NCT00840372
Title: Semi-blunt Needles: is Outcome Better?
Acronym: Needles
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Laura LABRIOLA, M.D., Cliniques Universitaires Saint-Luc, Université Catholique de Louvain
Other Study IDs: Needles; Semi-blunt needles
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Hemodialysis Patients; Vascular Abord: Native Arterio-venous Fistula; Buttonhole Cannulation
Keywords: Blunt needles; Semi-blunt needles; Buttonhole cannulation method

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Chronic hemodialysis patients, native arterio-venous fistula
  Interventions: Procedure: Buttonhole cannulation with semi-blunt needles
- 2: Chronic hemodialysis patients, native arterio-venous fistula
  Interventions: Procedure: Buttonhole cannulation with semi-blunt needles

INTERVENTIONS:
Procedure: Buttonhole cannulation with semi-blunt needles — Use of semi-blunt needles, compared to blunt needles, at every dialysis session

SUMMARY:
The aim of this observational study in patients chronically hemodialyzed by a native arterio-venous fistula is to determine the impact of the use of semi-blunt needles on the quality of the punction. The investigators have observed that cannulation with blunt needles (button-hole method) is sometimes difficult and the use of a sharp needle may be necessary, with consequently more hematomes and infections. Our hypothesis is that canulation with semi-blunt needles would be easier than with classical blunt needles, and consequently the use of sharp needles would become less frequent.

Inclusion criteria and study design are detailed below.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients
* Aged 18 years or more
* Dialyzed by a native arterio-venous fistula
* Cannuled by buttonhole method with blunt needles

Exclusion Criteria:

* Acute hemodialysis
* Puncture with 14G needles
* Puncture with a sole needle
* Arterio-venous grafts
* Patients transferred from another centre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hemodialysis patients dialyzed in Cliniques Universitaires Saint-Luc by a native arterio-venous fistula
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Incidence of AVF hematomes | Two months
Incidence of use of sharp needles | Two months

SECONDARY OUTCOMES:
Incidence of trampoline-effect | Two months
Incidence of AVF infections | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Labriola, M.D., Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium